CLINICAL TRIAL: NCT00532467
Title: Phase I, Double-Blind, Placebo-Controlled, Multiple Ascending Dose, Safety, Tolerability, Pharmacokinetic Study of SRX251 Capsules in Healthy Volunteers
Brief Title: Multiple Dose Safety Study of SRX251 Capsules in Healthy Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Azevan Pharmaceuticals (Industry)
Responsible Party: Eve Damiano, Sr. Vice President, Operations
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AVN002
Record Dates: First submitted 2007-09-18; First posted 2007-09-20 (Estimated); Last update posted 2008-03-13 (Estimated); Status verified 2008-03

CONDITIONS: Healthy
Keywords: healthy volunteers

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: SRX251

SUMMARY:
This study is the second study to evaluate SRX251 in healthy volunteers and it represents the first multiple dose study. The primary objective of this study is to evaluate the safety and tolerability of escalating multiple oral doses of SRX251 capsules for 5 days in healthy adult volunteers. Levels of the drug in blood plasma will also be determined.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy subjects between the ages of 18 and 55 years, inclusive. Subjects will be males or non-pregnant, non lactating females of non-childbearing potential.
2. Body mass index (BMI) of 18.5 to 34.0 kg/m2, inclusive, and a total body weight of >50kg (110 pounds).
3. In good health as determined by medical history, a baseline physical examination, vital signs, clinical laboratory tests and electrocardiogram (ECG) measurement.
4. Subject is willing and able to sign written informed consent prior to beginning study procedures.
5. Subject is willing and able to follow instructions, comply with the protocol requirements and make all required study visits.

Exclusion Criteria:

1. Evidence or history of clinically significant hematological, renal, endocrine, pulmonary, gastrointestinal, cardiovascular, hepatic, psychiatric, neurologic, or allergic disease (including drug allergies, but not excluding untreated, asymptomatic, seasonal allergies at time of dosing).
2. Pregnant or lactating females, or females of childbearing potential, defined as females who are not postmenopausal (postmenopausal females are defined as females who are 45 to 55 years of age and must be amenorrheic for at least 1 year PLUS have a serum FSH level within the laboratory's reference range for postmenopausal women) and females who have not had a hysterectomy and/or bilateral oophorectomy and/or tubal ligation.
3. Male subjects not willing to either abstain from sexual intercourse, or use one of the following methods of contraception from the first dose of trial medication until completion of follow-up procedures. Male subjects, without a vasectomy, must use a condom and be instructed that their female partner should use another form of contraception such as an IUD, spermicidal foam/gel/film/cream/suppository, diaphragm with spermicide, oral contraceptive, injectable progesterone, subdermal implant or a tubal ligation if the female partner could become pregnant from the time of the first dose of trial medication until completion of follow-up procedures.
4. Subject is positive for HIV, hepatitis B surface antigen or hepatitis C antibody tests at screening.
5. A general medical or psychological condition or behavior, including current substance dependence or abuse that, in the opinion of the investigator, might not permit the subject to complete the study or sign the informed consent.
6. Any other condition or clinically significant abnormal findings on the physical examination, medical history, or clinical laboratory results during screening that, in the opinion of the Principal Investigator, would make the subject unsuitable for the study or put them at additional risk.
7. Inability to understand or follow study instructions.
8. Known allergy or hypersensitivity to the investigational study drug/placebo components.
9. Treatment with an investigational drug within 30 days preceding the first does of study medication.
10. Blood donation of approximately 500 mL or more within 56 days prior to dosing.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 50 (Actual)
Dates: Start 2007-09; Primary Completion 2008-02 (Actual); Study Completion 2008-02 (Actual)

PRIMARY OUTCOMES:
safety and tolerability | duration of protocol

SECONDARY OUTCOMES:
pharmacokinetics | according to protocol

CONTACTS AND LOCATIONS:
Overall Officials: Benno G Roesch, MD, Principal Investigator — Advanced Biomedical Research, Inc.
Locations (1):
- Advanced Biomedical Research, Inc., Hackensack, New Jersey, United States